CLINICAL TRIAL: NCT01748565
Title: Gastrin-Releasing Peptide and Bronchopulmonary Dysplasia
Acronym: GRP
Status: Completed | Type: Observational
Sponsor: Duke University (Other)
Collaborators: Indiana University (Other); University of North Carolina, Chapel Hill (Other)
Responsible Party: Sponsor
Other Study IDs: Pro00025462
Record Dates: First submitted 2012-10-29; First posted 2012-12-12 (Estimated); Last update posted 2024-04-12 (Actual); Status verified 2016-08

CONDITIONS: Bronchopulmonary Dysplasia; Prematurity
Keywords: biomarkers; oxidative stress; BPD; prematurity
MeSH Terms: conditions — Bronchopulmonary Dysplasia; Premature Birth

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — urine specimens and saliva with DNA
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- premature infants: Infants born prematurely between 23-0/7 and 27-6/7 weeks post-menstrual age with and without bronchopulmonary dysplasia

SUMMARY:
The purpose of this study is to identify biological markers that might predict premature infants who are at a higher risk for developing BPD, and to correlate the presence of these markers with infant symptoms and lung function in the first year after discharge from the hospital.

DETAILED DESCRIPTION:
Bronchopulmonary dysplasia (BPD) is a common form of lung injury that can be triggered by premature birth and the unavoidable exposures to treatments regularly used for premature infants,including mechanical ventilation and oxygen as well as conditions that occur frequently among premature infants including infection. Almost all infants who are born prematurely are exposed to either mechanical ventilation, extra oxygen, and many will develop at least one infection; however, not all premature infants will develop BPD. There is currently no way to identify those infants who are at risk for developing BPD, nor are there prognostic or diagnostic tests to determine the severity of lung disease in the first year after discharge from the hospital.

The application of UPLC-tandem mass spectrometry for quantification of urinary biomarkers of oxidative stress is an important technical innovation that will permit sensitive and reproducible analyses of urinary biomarkers with minimal sample preparation to better define disease phenotypes. Establishing a direct correlation between biomarkers of oxidative stress and GRP will accelerate investigation into the mechanisms leading to chronic pediatric lung disease and childhood origins of pulmonary disease.

ELIGIBILITY:
Inclusion Criteria:

* Gestational age at birth 23-0/7 to 27-6/7 weeks post-menstrual age

Exclusion Criteria:

* Are not considered to be viable (decision made not to provide life-saving therapies)
* Have congenital heart disease (not including PDA and hemodynamically insignificant VSD or ASD)
* Have structural abnormalities of the upper airway, lungs or chest wall
* Have other congenital malformations or syndromes that adversely affect life expectancy or cardio-pulmonary development
* Unlikely to return to the clinic for follow-up visits

Max Age: 7 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Patients in the neonatal intensive care unit at Duke Medical Center or Riley Children's Hospital
Sampling Method: Non-Probability Sample
Enrollment: 260 (Actual)
Dates: Start 2012-05; Primary Completion 2016-08 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
urine GRP levels | day-of-life 1-4
  Comparing urine GRP levels to urine biomarkers of oxidative stress in infants with and without BPD
urine GRP levels | 36 weeks post-menstrual age
  Comparing urine GRP levels to urine biomarkers of oxidative stress in infants with and without BPD
urine GRP levels | 4-6 months corrected age
  Comparing urine GRP levels to urine biomarkers of oxidative stress in infants with and without BPD
urine GRP levels | 12-14 months corrected age
  Comparing urine GRP levels to urine biomarkers of oxidative stress in infants with and without BPD
infant pulmonary function tests | 4-6 months corrected age
  The association of urine GRP levels and the severity of lung disease as determined by pulmonary function tests in infants with and without BPD
infant pulmonary function tests | 12-14 months corrected age
  The association of urine GRP levels and the severity of lung disease as determined by pulmonary function tests in infants with and without BPD

CONTACTS AND LOCATIONS:
Overall Officials: Charles M Cotten, MD, Principal Investigator — Duke University
Locations (2):
- United States (2):
  - Riley Children's Hospital, Indianapolis, Indiana
  - Duke University Medical Center, Durham, North Carolina